CLINICAL TRIAL: NCT03186352
Title: Clinical Effect of Photoactivated Disinfection on Primary Root Carious Lesions After Partial Caries Removal
Acronym: PAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: WarsawMUKB/32/2016/1
Record Dates: First submitted 2017-06-12; First posted 2017-06-14 (Actual); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Primary Root Caries
Keywords: photodynamic therapy; photoactivated disinfection; primary root caries lesion; cavity disinfection; lasers; root caries
MeSH Terms: conditions — Root Caries | interventions — Photochemotherapy

STUDY DESIGN:
Intervention Model Description: Sample for microbiological evaluation is to be taken from each patient before and after intervention (PAD). Before-After Study Type.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- after intervention (Experimental): sample for microbial analysis it taken with sterile a rose bur (size 014) on micro motor after intervention
  Interventions: Procedure: photoactivated disinfection

INTERVENTIONS:
Procedure: photoactivated disinfection — After manual preparation of the cavity with an excavator and taking a sample for a microbial analysis with a rose bur on micro motor (size 014) the cavity undergoes the procedure of photodynamic disinfection:
  application of photosensitizer 'Fotosan' Agent (CMS Dental, Denmark) for 5 minutes, radiation with low power laser, wavelength 635 nm power 200mW 120 s. ('Lasotronix', DiodeLX model SMART) rinsing with water and drying
  Other Names: Photodynamic therapy; photodynamic antimicrobial chemotherapy

SUMMARY:
The problem of root caries has been increasing in last decades as the an average life expectancy is rising. Due to progress of medicine and dentistry humans also maintain natural dentition longer.

The aim of the study is to determine the effectiveness of photoactivated disinfection / photodynamic therapy / photodynamic antimicrobial therapy in elimination of cariogenic bacteria after manual root caries removal.

If proved to be effective in eliminating bacteria from prepared cavity PAD could be incorporated in the protocol of treatment of root cavities.

DETAILED DESCRIPTION:
Elimination of cariogenic bacteria is to be determined in this study - Mutans streptococci, Lactobacillus spp. and Actinomyces spp.

After manual preparation of the cavity with an excavator and taking a sample for a microbial analysis with a rose bur on micro motor (size 014) the cavity undergoes the procedure of photodynamic disinfection:

* application of photosensitizer 'Fotosan Agent' (CMS Dental, Denmark) for 5 minutes,
* radiation with low power laser, wavelength 635 nm power 200mW 120 s. ('Lasotronix', DiodeLX model SMART)
* rinsing with water and drying

After photodynamic disinfection another sample for microbial analysis is taken form the neighboring area to get the material for a comparison analysis.

Filling the cavity with a material for permanent fillings (glass-ionomer cement)

Samples are inoculated on:

* Mitis-Salivarius ('Difco') for Streptococci
* Rogosa SL 2% aqar ('Oxoid') for Lactobacillus
* Columbia with blood for Actinomyces (2 dilutions - 1:10 and 1:100)

ELIGIBILITY:
Inclusion Criteria:

* more than 10 teeth
* at least one tooth with primary caries lesion with contraindicated non-invasive treatment (lesion which needs to be prepared and filled with material for permanent fillings); tooth with no clinical and/or radiological symptoms of pulp involvement.
* no systemic disease

Exclusion Criteria:

* systemic diseases (may affect saliva flow and properties)
* antibiotic therapy in previous 3 months before the appointment

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-07-11 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-02-28 (Estimated)

PRIMARY OUTCOMES:
elimination of bacteria | 7 day
  determination of amount of Colony Forming Units per ml

CONTACTS AND LOCATIONS:
Locations (1):
- Zakład Stomatologii Zachowawczej, Warsaw, Woj. Mazowieckie, Poland